CLINICAL TRIAL: NCT00815893
Title: Interventional Study of Dexmedetomidine for Sedating Anticipated Difficult Airway Patients Undergoing Awake Fiberoptic Nasal Intubation
Brief Title: The Feasibility of Dexmedetomidine for Awake Fiberoptic Nasal Intubation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Koung-Shing Chu, Department of Anesthesiology, Kaohsiung Medical University Chung-Ho Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMUHIRB-96-09-02
Record Dates: First submitted 2008-12-10; First posted 2008-12-31 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2008-12

CONDITIONS: Awake Fiberoptic Nasal Intubation
Keywords: Dexmedetomidine; Fiberoptic nasal intubation; satisfaction
MeSH Terms: conditions — Personal Satisfaction | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 dex group (Experimental): received dexmedetomidine (1.0 mcg/kg) infusion
  Interventions: Drug: dexmedetomidine
- 2 control group (Placebo Comparator): received 0.9% saline
  Interventions: Drug: Normal Saline 0.9%
- 3 Propofol group (Active Comparator): received 1% propofol using effect-site TCI(Base Primea, Fresenius, France)
  Interventions: Drug: propofol 1%

INTERVENTIONS:
Drug: dexmedetomidine — dexmedetomidine 1.0 mcg/kg infusion for 10minutes
  Other Names: Precedex 100microg/ml
  Arms: 1 dex group
Drug: Normal Saline 0.9% — 0.9% Normal Saline 0.25ml/kg infusion for 10minues
  Other Names: saline 0.9% Nacl
  Arms: 2 control group
Drug: propofol 1% — Propofol: The initial target = 3 μg/ml. The TCI is adjusted by 0.5μg/ml according to patient comfort during the procedure.
  The Orchestra® Base Primea(Fresenius, Brezins, France) offers a Target Controlled Infusion (TCI) target controlled infusion.
  Other Names: propofol
  Arms: 3 Propofol group

SUMMARY:
The objective of this study is to evaluate the feasibility of dexmedetomidine infusion for oral cancer patients undergoing awake fiberoptic nasal intubation. We hypothesized that a loading dose of intravenous dexmedetomidine before awake fiberoptic nasal intubation for oral cancer patients undergoing general anesthesia will provide adequate sedation and analgesia without respiratory depression and upper airway obstruction.

DETAILED DESCRIPTION:
Case number: 60, ASA I-III oral cancer patients with limited mouth opening

Patients will be randomly allocated into three groups, Dex group received dexmedetomidine (1.0 mcg/kg) infusion, Control group received saline, and Propofol group received 1% Propofol administrated usng effect-site TCI.

Main outcome was evaluated by grading scores presenting conditions for nasal intubation, post-intubation and satisfaction.

Other analysed parameters included airway obstruction, hemodynamic changes, treatment for hemodynamics response, consumption time for intubation, amnesia level, and postoperative adverse events. All outcome measurements were classified by scoring systems.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients with limited mouth opening
* Undergoing awake fiberoptic nasal intubation for elective surgery

Exclusion Criteria:

* a history of severe bradycardia
* any type of A-V block in EKG
* heart failure
* liver cirrhosis
* thrombocytopenia
* coagulopathy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
grading scores presenting conditions for nasal intubation | before and after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Koung-Shing Chu, Master, Study Director — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Hospital, Kaohsiung City, Taiwan